CLINICAL TRIAL: NCT00974480
Title: Single Blind Study to Evaluate the Tolerance and Effectiveness of Redermic Versus Rejuva-A™ (0.025% Tretinoin) and Redermic in Combination With Rejuva-A™ (0.025% Tretinoin) Under Normal Conditions in Subjects With Signs of Aging
Brief Title: Comparison of Redermic, Rejuva-A and Combination of Both Redermic and Rejuva-A in Subjects With Signs of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Principal Investigator, Robert BISSONNETTE, President and Dermatologist, Cosmetique Active International
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LRP09008
Record Dates: First submitted 2009-07-24; First posted 2009-09-10 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Skin Aging
Keywords: Skin; Aging; Rejuva-a; Redermic
MeSH Terms: interventions — Ascorbic Acid; Tretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Redermic (Experimental): Cream was applied twice a day every day, morning and evening for 24 weeks.
  Interventions: Other: Redermic
- Rejuva-A (Active Comparator): Week 1, Rejuva-A cream was applied to face in the evening twice a week. Weeks 2 & 3, Rejuva-A cream was applied to the face in the evening three times a week. Weeks 4-24, Rejuva-A cream was applied to the face in the evening every other day. In cases of intolerance, returned to the previous dosage and remained there until the end of study. Hydrating cream was applied to the face in the morning every day for 24 weeks.
  Interventions: Drug: Tretinoin (Rejuva-A)
- Combination of Redermic and Rejuva-A (Active Comparator): Week 1, Rejuva-A cream was applied to face in the evening twice a week. Weeks 2 & 3, Rejuva-A cream was applied to the face in the evening three times a week. Weeks 4-24, Rejuva-A cream was applied to the face in the evening every other day. In cases of intolerance, returned to the previous dosage and remained there until the end of study. Redermic was applied every evening when Rejuva-A™ was not applied, as well as every morning.
  Interventions: Other: Redermic; Drug: Tretinoin (Rejuva-A)

INTERVENTIONS:
Other: Redermic — Cosmetic cream formulation 609637 43.
  Other Names: madescassoside; vitamin C
  Arms: Combination of Redermic and Rejuva-A; Redermic
Drug: Tretinoin (Rejuva-A) — Tretinoin 0.025% cream.
  Other Names: Rejuva-A
  Arms: Combination of Redermic and Rejuva-A; Rejuva-A

SUMMARY:
Facial skin aging is a complex process combining factors such as sun exposure, smoking and those that are believed to be inherited. Changes in the skin over time including decreased thickness result in skin atrophy, wrinkling, sagging, yellowness and changes in pigmentation. Redermic is a cosmetic cream that has been evaluated clinically but not in comparison to tretinoin nor in combination with tretinoin. There is no data on the safety and efficacy of Redermic as compared to topical tretinoin.

Rejuva is a cream currently approved by Health Canada for the treatment of photodamaged skin. It contains 0.025% tretinoin one of the most widely studied topical product for skin aging. Studies have shown that topical tretinoin increases collagen synthesis and epidermal thickness thereby improving the appearance of skin aging. The efficacy of Rejuva combined with another topical cosmetic cream such as Redermic in the treatment of skin aging is unknown.

One hundred and twenty (120) subjects with signs of skin aging participated in this single-blind study to evaluate the efficacy and tolerance of Redermic versus Rejuva-A™ (0.025% tretinoin) and Redermic in combination with Rejuva-A™ (0.025% tretinoin).

DETAILED DESCRIPTION:
Facial skin aging is a complex and multifactorial process combining extrinsic and intrinsic factors. Major extrinsic factors include sun exposure and smoking while intrinsic factors are believed to be genetically programmed.

Changes in the dermis are responsible for many of the important clinical changes associated with skin aging. With age there is a decrease in the number of fibroblasts and a decrease in their ability to synthesize collagen which results in a decrease in collagen I and II. This is coupled with an increase in matrix metalloproteinases activity. Skin biopsies from elderly volunteers show changes in collagen bundles which become fragmented and disorganized as well as in elastin fibers which are decreased. Changes also occur in the epidermis including a decrease in epidermal thickness and a change in the morphology of keratinocytes of the basal layer. Clinically these changes result in skin atrophy, increased skin laxity, wrinkling, sagging, yellowness and changes in pigmentation.

Redermic is a cosmetic cream containing vitamin C and madecassoside. A preliminary 20 subject split face study has shown that this product was well tolerated and could improve signs of skin aging. To evaluate changes in skin aging this study used a clinical evaluation of the face, skin hydration, the fringe technique, skin biopsies and skin elasticity measurements. The investigators did not perform transepidermal water loss (TEWL), facial skin evaluation using a photonumeric guideline, evaluation of photoaging by panel of blinded dermatologists or skin replica evaluations. There is no data on the combination of Redermic with tretinoin or on the safety and efficacy of Redermic as compared to topical tretinoin.

Rejuva is a cream currently approved by Health Canada for the treatment of photodamaged skin. It contains 0.025% tretinoin one of the most widely studied topical product for skin aging. Studies have shown that topical tretinoin increases collagen synthesis and epidermal thickness thereby improving the appearance of skin aging. The efficacy of Rejuva combined with another topical cosmetic cream such as Redermic in the treatment of skin aging is unknown.

The main objective of this single-blind study was to assess efficacy of the anti aging effect and the tolerance of Redermic alone compared to Rejuva-A™ (0.025% tretinoin) alone or in combination with Rejuva-A™ (0.025% tretinoin).

One hundred and twenty (120) subjects with signs of skin aging participated in this single-blind study to evaluate the efficacy and tolerance of Redermic versus Rejuva-A™ (0.025% tretinoin) and Redermic in combination with Rejuva-A™ (0.025% tretinoin). Subjects were randomized (1:1:1) in three groups of forty (40), and were asked to apply study product to the face (except to eyelids, nostrils and other mucous membranes) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are female, between 45 and 55 years of age.
* Females of childbearing potential have had a negative urine pregnancy test prior to randomization.
* Subjects are willing to use adequate contraceptive method or are surgically sterile (including tubal ligation), post-menopausal, abstinent or with a same-sex partner. Adequate means of contraception include; intra-uterine device (IUD) in use for 30 days before Day 0, barrier methods and spermicide in use at least 14 days before Day 0 or oral contraceptive in use for at least 30 days before Day 0.
* Subjects are willing to avoid prolonged exposure to UV radiation for the duration of the study.
* Subjects are capable of giving written informed consent.
* Subjects have changes associated with facial skin aging/photodamaged skin.

Exclusion Criteria:

* Subjects are male.
* Subjects are pregnant or lactating.
* Subjects have a known allergy to Redermic, Rejuva-A™ or to any component of the tested products.
* Subjects have made use of tretinoin, adapalene, tazarotene or other topical medications for the treatment of facial skin aging during the 12 weeks preceding Day 0.
* Subjects have applied topical alpha hydroxyl acids within 28 days of Day 0.
* Subjects have used or plan to use systemic corticosteroids within 28 days of Day 0 or during the study.
* Subjects have made use of a non-medication topical product directed at improving skin aging during the 28 days preceding Day 0.
* Subjects have a hypersensitivity to any retinoids.
* Subjects have a history of alcohol or drug abuse in the past year.
* Subjects are participating in another interventional study.
* Subjects have had a previous intense pulsed light treatment to the face.
* Subjects have had a previous laser treatment to the face directed at improving skin aging.
* Subjects have the presence of skin diseases such as psoriasis or dermatitis on the face that could interfere with study evaluations.
* Planned or unavoidable exposure to intense ultraviolet (UV) radiation during the study (such as sun tanning salons, vacations in a sunny climate or outdoor worker).
* Subjects have had a botulinum toxin A injection treatment on the face within 2 years of Day 0 or plan to receive this treatment during the study.
* Subjects have had a filler injection (collagen, hyaluronic acid, etc..) on the face within 2 years of Day 0 or plan to receive this treatment during the study.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from September 2009 to January 2010 at a research clinic.
Groups:
- Redermic: Cream applied twice a day every day, morning and evening for 24 weeks.
- Rejuva-A: Week 1, Rejuva-A cream was applied to face in the evening twice a week. Weeks 2 & 3, Rejuva-A cream was applied to the face in the evening three times a week. Weeks 4-24, Rejuva-A cream was applied to the face in the evening every other day. In cases of intolerance, subjects returned to the previous dosage and remained there until the end of study. Neutral cream was applied to the face in the morning every day for 24 weeks.
- Combination of Redermic and Rejuva-A: Week 1, Rejuva-A cream was applied to face in the evening twice a week. Weeks 2 & 3, Rejuva-A cream was applied to the face in the evening three times a week. Weeks 4-24, Rejuva-A cream was applied to the face in the evening every other day. In cases of intolerance, subjects returned to the previous dosage and remain there until the end of study. Redermic was applied every evening when Rejuva-A™ was not applied, as well as every morning.
Period: Overall Study
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Started | 40 | 40 | 40
Completed | 29 | 33 | 30
Not Completed | 11 | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 40 | 120
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.85 (3.18) | 51.15 (3.20) | 50.53 (2.84) | 50.51 (3.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 40 | 120
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 40 | 40 | 120
Skin aging measured with photonumeric scale [Mean (Standard Deviation); unit: Units on a Scale] — Scoring was accomplished by matching each part of the face (forehead, glabella, corners of the mouth, nasal labial fold, crow's feet, below eyes and upper lip) to photographs in the scales and reporting the appropriate number in the tables. All individual scores were added to obtain the total score (Less signs of skin aging = 0, more signs of skin aging = 41.6).
  Units on a Scale | 22.23 (7.10) | 21.88 (5.83) | 22.14 (5.13) | 22.08 (6.06)
Transepidermal water loss (TEWL) [Mean (Standard Deviation); unit: g / m² / h] — Trans Epidermal Water Loss (TEWL) was measured with a DermaLab device (Cortex Technology, Denmark) equipped with a TEWL probe. Measurements were performed with the subject lying down on the back in a room with controlled temperature (20°C +/-2) and relative humidity (45% +/- 15%). All measurements were performed at least 30 minutes after the subject was transferred into this room. The measurements were performed on the cheek. Care was taken to use the same cheek for each subject throughout the study.
  g / m² / h | 9.90 (3.32) | 9.61 (2.95) | 9.71 (2.47) | 9.74 (2.91)
Skin hydration (conductance) [Mean (Standard Deviation); unit: µsiemens (µmho)] — Skin hydration was measured with a DermaLab device (Cortex Technology, Denmark) equipped with a skin hydration probe.
  Measurements were performed in a room with controlled temperature (20°C +/-2) and humidity (45% +/- 15%). All measurements were performed at least 30 minutes after the subject had been transferred into this room. Care was taken to use the same cheek for each subject throughout the study. Higher values indicate greater hydration.
  µsiemens (µmho) | 51.00 (25.58) | 64.35 (42.44) | 57.25 (26.54) | 57.53 (32.64)
Skin elasticity [Mean (Standard Deviation); unit: kilo Pascals] — Skin elasticity was measured with a DermaLab device (Cortex Technology, Denmark) equipped with a skin elasticity probe. Pressure required to raise the skin 1mm was recorded. Measurements were performed on the upper cheeks and care was taken to use the same location for all measurements. Final measurements were the average of left and right cheeks. When the product is a moisturizer, lower pressures are indicative of efficacy.
  kilo Pascals | 20.61 (10.83) | 19.27 (8.51) | 20.61 (9.75) | 20.16 (9.68)
Crow's feet replicas - area ratio [Mean (Standard Deviation); unit: mm²] — An illuminator is used to cross illuminate the specimen (silicone mold replicas) perpendicular to the major lines which accentuate the surface details. The resulting image which consists of a series of shadows that directly correspond to the pattern of wrinkles is digitized for analysis. One can measure changes in skin surface topography by selecting an area range (shadow size) that allows one to directly determine the projected area of the shadowed region associated with the wrinkles and major lines. The Area Ratio is the area of the shadows. The higher the ratio, the greater the wrinkling.
  mm² | 7.98 (6.31) | 5.87 (4.78) | 9.28 (7.71) | 7.53 (5.52)
Clinical skin evaluation [Mean (Standard Deviation); unit: Units on a scale] — A clinical skin evaluation of the face was performed by a dermatologist using 8 scales (skin hydration, radiance, roughness, spots, laxity, skin tone homogeneity, softness, relief (variations in depth)). The individual scores were totalled (worst = 0, best = 47) and the total score was used for analyses.
  Units on a scale | 29.05 (5.52) | 29.20 (5.96) | 28.65 (6.06) | 28.97 (5.81)
Sensitivity of the face evaluated by subject [Mean (Standard Deviation); unit: Units on a scale] — Sensitivity of the entire face evaluated by the subject was performed using 4 different 10 cm visual analog scales (pruritus, tingling, burning, tightness). Each score was analysed separately.
  Each score is from 0 = absent to 10 important.
  Units on a scale
    Pruritus | 0.94 (1.51) | 1.01 (1.88) | 0.65 (1.73) | 0.87 (1.71)
    Tingling | 0.99 (1.51) | 0.69 (1.28) | 1.04 (1.77) | 0.91 (1.53)
    Burning | 0.83 (1.67) | 0.55 (1.27) | 0.45 (1.19) | 0.61 (1.39)
    Tightness | 1.56 (2.02) | 1.62 (2.21) | 1.30 (2.47) | 1.49 (2.23)
Facial skin self-evaluation [Mean (Standard Deviation); unit: Units on a scale] — A visual analog scale of 13 evaluations were performed by the subject. Scale is from 1 - 10 for each evaluation individually evaluated. 0 = absent, 10 = important
  Units on a scale
    Hydration | 4.65 (2.01) | 4.61 (1.81) | 4.98 (1.55) | 4.75 (1.79)
    Firmness | 4.67 (2.00) | 5.34 (2.27) | 4.62 (1.60) | 4.88 (1.99)
    Radiance | 5.14 (1.72) | 4.86 (1.69) | 5.01 (2.10) | 5.00 (1.83)
    Softness | 5.54 (1.54) | 5.10 (2.19) | 5.24 (1.93) | 5.29 (1.90)
    Comfort | 5.39 (1.97) | 5.75 (1.93) | 6.31 (2.48) | 5.82 (2.16)
    Smoothness | 6.20 (2.02) | 6.53 (2.25) | 6.51 (1.95) | 6.41 (2.07)
    Fine Lines | 5.06 (1.85) | 5.52 (2.12) | 5.11 (2.12) | 5.23 (2.03)
    Wrinkles | 5.14 (2.14) | 5.67 (2.15) | 5.06 (2.17) | 5.29 (2.15)
    Spots | 2.92 (2.31) | 3.97 (2.60) | 4.17 (2.81) | 3.68 (2.62)
    Roughness | 2.65 (2.14) | 3.02 (2.62) | 2.50 (2.14) | 2.72 (2.31)
    Imperfections | 4.73 (2.41) | 5.08 (2.18) | 5.24 (2.57) | 5.01 (2.38)
    Dryness | 5.01 (2.32) | 5.15 (2.34) | 4.35 (2.65) | 4.83 (2.45)
    Redness | 3.04 (2.65) | 3.00 (3.09) | 2.92 (3.00) | 2.99 (2.89)
Tolerance evaluated by investigator [Mean (Standard Deviation); unit: Units on a scale] — Tolerance was studied by evaluating scaling, dryness, erythema and burning/itching sensation on a 5-point scale.
  Scaling, Dryness and Erythema Evaluations
  - None (0) - Very Severe = (4)
  Burning and Itching Evaluation Scale
  * None (0) = Normal, no discomfort
  * Mild (1) = Slight discomfort that is not bothersome
  * Moderate (2) = Discomfort that is somewhat bothersome
  * Marked (3) = Discomfort that is bothersome and that occasionally interferes with normal daily activities
  * Severe (4) = Continuous discomfort that interferes with normal daily activities
  Units on a scale
    Scaling | 0.08 (0.27) | 0.05 (0.22) | 0.03 (0.16) | 0.05 (0.22)
    Dryness | 0.13 (0.33) | 0.10 (0.30) | 0.15 (0.36) | 0.13 (0.33)
    Erythema | 0.05 (0.32) | 0.0 (0.0) | 0.08 (0.27) | 0.04 (0.24)
    Burning and itching | 0.13 (0.33) | 0.18 (0.59) | 0.08 (0.27) | 0.13 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Skin Aging Measured With the Photonumeric Scale.
Description: Scoring was accomplished by matching each part of the face (forehead, glabella, corners of the mouth, nasal labial fold, crow's feet, below eyes and upper lip) to photographs in the scales and reporting the appropriate number in the tables. All individual scores were added to obtain the total score (Less signs of skin aging = 0, more signs of skin aging = 41.6).
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
Units on a scale
  Week 12 | 21.25 (6.60) | 21.36 (5.93) | 21.21 (5.29)
  Week 24 | 21.03 (6.81) | 20.92 (5.75) | 21.31 (5.26)

2. Secondary Outcome: Photographic Evaluation by a Panel of Blinded Dermatologists.
Description: A blinded panel of two dermatologists had to identify independently which of the two photographs had an improvement or if there was no noticeable difference between them. The two photographs of each subject were randomized to keep the blind.
  When the Week 24 photograph was selected as the one showing an improvement, it was scored by the statistician as "improvement". When the Day 0 photograph was selected as the one showing an improvement, it was scored by the statistician as "worsening". When there was no noticeable difference between the photographs, it was scored as "stable".
Time Frame: 24 weeks
Population: Analysis was intent to treat (ITT). Photographs taken at early termination visit were not available for every early termination subject as some subjects refused to have their photographs taken. Thus, early termination and lost to follow-up subjects were excluded from this analysis. The total number of subjects included in the ITT analysis was 92.
Measure: Number; unit: Participants
Groups:
- Redermic - Assessor 1; Redermic - Assessor 2: Cream applied twice a day every day, morning and evening for 24 weeks.
- Rejuva-A - Assessor 1; Rejuva-A - Assessor 2: Week 1, Rejuva-A cream was applied to face in the evening twice a week. Weeks 2 & 3, Rejuva-A cream was applied to the face in the evening three times a week. Weeks 4-24, Rejuva-A cream was applied to the face in the evening every other day. In cases of intolerance, subjects returned to the previous dosage and remained there until the end of study. Neutral cream was applied to the face in the morning every day for 24 weeks.
- Combination of Redermic and Rejuva-A - Assessor 1; Combination of Redermic and Rejuva-A - Assessor 2: Week 1, Rejuva-A cream was applied to face in the evening twice a week. Weeks 2 & 3, Rejuva-A cream was applied to the face in the evening three times a week. Weeks 4-24, Rejuva-A cream was applied to the face in the evening every other day. In cases of intolerance, subjects returned to the previous dosage and remained there until the end of study. Redermic was applied every evening when Rejuva-A™ was not applied, as well as every morning.
Arm/Group | Redermic - Assessor 1 | Rejuva-A - Assessor 1 | Combination of Redermic and Rejuva-A - Assessor 1 | Redermic - Assessor 2 | Rejuva-A - Assessor 2 | Combination of Redermic and Rejuva-A - Assessor 2
Number analyzed (Participants) | 29 | 33 | 30 | 29 | 33 | 30
Participants
  Worsening | 7 | 4 | 5 | 5 | 4 | 1
  Stable | 14 | 19 | 18 | 19 | 21 | 23
  Improvement | 8 | 10 | 7 | 5 | 8 | 6

3. Secondary Outcome: Trans-epidermal Water Loss (TEWL).
Description: Trans Epidermal Water Loss (TEWL) was measured with a DermaLab device (Cortex Technology, Denmark) equipped with a TEWL probe. Measurements were performed with the subject lying down on the back in a room with controlled temperature (20°C +/-2) and relative humidity (45% +/- 15%). All measurements were performed at least 30 minutes after the subject was transferred into this room. The measurements were performed on the cheek. Care was taken to use the same cheek for each subject throughout the study.
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: g / m² / h
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
g / m² / h
  Week 12 | 10.51 (3.45) | 12.33 (4.39) | 13.12 (5.72)
  Week 24 | 10.20 (3.12) | 12.64 (4.47) | 12.45 (6.00)

4. Secondary Outcome: Skin Hydration (Conductance)
Description: Skin hydration was measured with a DermaLab device (Cortex Technology, Denmark) equipped with a skin hydration probe.
  Measurements were performed in a room with controlled temperature (20°C +/-2) and humidity (45% +/- 15%). All measurements were performed at least 30 minutes after the subject had been transferred into this room. Care was taken to use the same cheek for each subject throughout the study. Higher values indicate greater hydration.
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: µsiemens (µmho)
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
µsiemens (µmho)
  Week 12 | 65.10 (34.38) | 84.25 (51.14) | 74.85 (37.56)
  Week 24 | 66.45 (30.48) | 83.65 (47.59) | 80.70 (45.80)

5. Secondary Outcome: Skin Elasticity.
Description: Skin elasticity was measured with a DermaLab device (Cortex Technology, Denmark) equipped with a skin elasticity probe. Pressure required to raise the skin 1mm was recorded. Measurements were performed on the upper cheeks and care was taken to use the same location for all measurements. Final measurements were the average of left and right cheeks. When the product is a moisturizer, lower pressures are indicative of efficacy.
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: kilo Pascals
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
kilo Pascals
  Week 12 | 19.56 (11.09) | 18.16 (10.65) | 17.34 (7.99)
  Week 24 | 20.30 (10.54) | 17.21 (9.42) | 18.30 (9.19)

6. Secondary Outcome: Area Ratio - Analysis of Skin Replicas of Crow's Feet.
Description: An illuminator is used to cross illuminate the specimen (silicone mold replicas) perpendicular to the major lines which accentuate the surface details. The resulting image which consists of a series of shadows that directly correspond to the pattern of wrinkles is digitized for analysis. One can measure changes in skin surface topography by selecting an area range (shadow size) that allows one to directly determine the projected area of the shadowed region associated with the wrinkles and major lines. The Area Ratio is the area of the shadows. The higher the ratio, the greater the wrinkling.
Time Frame: 24 weeks
Population: Only the per protocol (PP) population was considered for this analysis. Early termination and lost subjects were excluded from this analysis. Furthermore, some replicas of subjects who completed the study could not be analyzed with precision and were consequently excluded from the analysis by the laboratory.
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 21 | 21 | 28
mm² | 6.35 (5.49) | 3.52 (2.99) | 7.35 (6.38)

7. Secondary Outcome: Clinical Skin Evaluation.
Description: A clinical skin evaluation of the face was performed by a dermatologist using 8 scales (skin hydration, radiance, roughness, spots, laxity, skin tone homogeneity, softness, relief (variations in depth)). The individual scores were totalled (worst = 0, best = 47) and the total score was used for analyses.
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
Units on a scale
  Week 12 | 29.90 (4.66) | 30.35 (5.14) | 29.63 (5.06)
  Week 24 | 31.00 (4.89) | 30.90 (5.51) | 30.25 (4.74)

8. Secondary Outcome: Sensitivity of the Face Evaluated by Subject.
Description: Sensitivity of the entire face evaluated by the subject was performed using 4 different 10 cm visual analog scales (pruritus, tingling, burning, tightness). Each score was analysed separately.
  Each score is from 0 = absent to 10 important.
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
Units on a scale
  Pruritus sensation Week 12 | 1.13 (2.06) | 1.62 (2.31) | 1.95 (2.69)
  Pruritus sensation Week 24 | 1.01 (1.77) | 1.79 (2.06) | 2.06 (2.78)
  Tingling sensation Week 12 | 1.36 (2.41) | 2.02 (2.50) | 3.06 (3.08)
  Tingling sensation Week 24 | 0.85 (1.44) | 2.24 (2.53) | 2.33 (2.98)
  Burning sensation Week 12 | 1.34 (2.37) | 2.61 (2.84) | 3.55 (3.36)
  Burning sensation Week 24 | 0.69 (1.64) | 1.89 (2.59) | 2.85 (3.41)
  Tightness sensatioin Week 12 | 1.57 (2.20) | 1.94 (2.21) | 3.00 (3.10)
  Tightness sensation Week 24 | 1.45 (2.00) | 2.45 (2.94) | 2.27 (2.56)

9. Secondary Outcome: Facial Skin Self-evaluation.
Description: A visual analog scale of 13 evaluations were performed by the subject. Scale is from 1 - 10 for each evaluation individually evaluated. 0 = absent, 10 = important.
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
Units on a scale
  Hydration Week 12 | 6.01 (2.08) | 5.54 (2.02) | 5.53 (2.32)
  Hydration Week 24 | 6.80 (2.14) | 6.12 (2.18) | 5.93 (1.90)
  Firmness Week 12 | 5.43 (2.12) | 5.10 (2.32) | 5.24 (1.91)
  Firmness Week 24 | 5.72 (2.23) | 5.60 (1.92) | 5.59 (1.64)
  Radiance Week 12 | 5.63 (1.63) | 5.41 (2.12) | 5.76 (1.91)
  Radiance Week 24 | 6.11 (1.91) | 5.81 (1.74) | 6.07 (1.80)
  Softness Week 12 | 6.20 (1.84) | 5.53 (1.84) | 5.80 (1.47)
  Softness Week 24 | 6.40 (2.12) | 5.60 (2.06) | 6.18 (1.70)
  Comfort Week 12 | 6.29 (2.16) | 6.21 (1.89) | 5.96 (2.16)
  Comfort Week 24 | 7.05 (2.01) | 6.20 (2.23) | 6.49 (1.84)
  Smoothness Week 12 | 6.83 (1.80) | 6.88 (2.16) | 6.63 (1.81)
  Smoothness Week 24 | 7.26 (1.81) | 6.98 (1.93) | 6.85 (1.95)
  Fine lines Week 12 | 5.15 (1.85) | 4.82 (2.02) | 5.18 (2.40)
  Fine lines Week 24 | 5.00 (2.01) | 5.03 (2.02) | 4.97 (2.38)
  Wrinkles Week 12 | 4.99 (2.07) | 5.06 (2.08) | 5.38 (2.27)
  Wrinkles Week 24 | 5.43 (2.14) | 5.40 (2.23) | 5.23 (1.89)
  Spots Week 12 | 3.13 (2.29) | 4.32 (2.77) | 4.00 (2.62)
  Spots Week 24 | 3.22 (2.65) | 4.35 (2.95) | 3.57 (2.69)
  Roughness Week 12 | 2.74 (2.05) | 3.44 (2.64) | 3.41 (2.32)
  Roughness Week 24 | 2.96 (2.60) | 3.09 (2.75) | 3.49 (2.38)
  Imperfections Week 12 | 4.52 (2.30) | 4.39 (2.23) | 4.73 (2.80)
  Imperfections Week 24 | 4.27 (2.56) | 4.82 (2.33) | 4.58 (2.51)
  Dryness Week 12 | 4.21 (2.59) | 4.30 (2.71) | 4.60 (2.87)
  Dryness Week 24 | 3.72 (2.52) | 4.21 (2.82) | 4.66 (2.75)
  Redness Week 12 | 3.33 (3.10) | 3.94 (2.66) | 3.75 (2.81)
  Redness Week 24 | 3.16 (2.68) | 3.51 (2.80) | 3.96 (3.11)

10. Secondary Outcome: Tolerance Evaluated by Investigator.
Description: Tolerance was studied by evaluating scaling, dryness, erythema and burning/itching sensation on a 5-point scale.
  Scaling, Dryness and Erythema Evaluations
  - None (0) - Very Severe = (4)
  Burning and Itching Evaluation Scale
  * None (0) = Normal, no discomfort
  * Mild (1) = Slight discomfort that is not bothersome
  * Moderate (2) = Discomfort that is somewhat bothersome
  * Marked (3) = Discomfort that is bothersome and that occasionally interferes with normal daily activities
  * Severe (4) = Continuous discomfort that interferes with normal daily activities
Time Frame: 12, 24 weeks
Population: Analysis was intent to treat (ITT) with Last Observation Carried Forward (LOCF) imputation technique.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Number analyzed (Participants) | 40 | 40 | 40
Units on a scale
  Scaling Week 12 | 0.10 (0.30) | 0.28 (0.55) | 0.15 (0.43)
  Scaling Week 24 | 0.10 (0.30) | 0.30 (0.56) | 0.33 (0.66)
  Dryness Week 12 | 0.15 (0.36) | 0.30 (0.52) | 0.23 (0.58)
  Dryness Week 24 | 0.13 (0.33) | 0.25 (0.49) | 0.35 (0.70)
  Erythema Week 12 | 0.15 (0.43) | 0.05 (0.22) | 0.10 (0.30)
  Erythema Week 24 | 0.13 (0.33) | 0.10 (0.30) | 0.23 (0.48)
  Burning and itching Week 12 | 0.03 (0.16) | 0.23 (0.58) | 0.23 (0.48)
  Burning and itching Week 24 | 0.03 (0.16) | 0.25 (0.67) | 0.23 (0.53)

ADVERSE EVENTS:
Arm/Group | Redermic | Rejuva-A | Combination of Redermic and Rejuva-A
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 3/40 | 10/40 | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Redermic (N=40) | Rejuva-A (N=40) | Combination of Redermic and Rejuva-A (N=40)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Redermic (N=40) | Rejuva-A (N=40) | Combination of Redermic and Rejuva-A (N=40)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Common Cold (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No